CLINICAL TRIAL: NCT02362438
Title: A Phase I Study of Intrathecal Administration of scAAV9/JeT-GAN for the Treatment of Giant Axonal Neuropathy
Brief Title: Intrathecal Administration of scAAV9/JeT-GAN for the Treatment of Giant Axonal Neuropathy
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 150073; 15-N-0073
Record Dates: First submitted 2015-02-12; First posted 2015-02-13 (Estimated); Last update posted 2026-01-05 (Actual); Status verified 2025-08-22

CONDITIONS: Giant Axonal Neuropathy; Gene Transfer
Keywords: Intrathecal; AAV9 Mediated Gene Transfer; Phase I; Safety Study; Giant Axonal Neuropathy
MeSH Terms: conditions — Giant Axonal Neuropathy

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- 10X (Experimental): Highest dose in the escalation scheme
  Interventions: Genetic: scAAv9/JeT-GAN
- 1X (Experimental): Lowest dose in the escalation scheme
  Interventions: Genetic: scAAv9/JeT-GAN
- 3.3X (Experimental): 2nd dose increase in escalation scheme
  Interventions: Genetic: scAAv9/JeT-GAN
- 5X (Experimental): 3rd dose increase in escalation scheme
  Interventions: Genetic: scAAv9/JeT-GAN

INTERVENTIONS:
Genetic: scAAv9/JeT-GAN — scAAV9/JeT-GAN is a biological gene transfer reagent

SUMMARY:
Title: Intrathecal Administration of scAAV9/JeT-GAN for the Treatment of Giant Axonal Neuropathy

Background:

- The Gigaxonin gene lets the body make a protein chemical called Gigaxonin. Nerves need Gigaxonin to work properly. Giant Axonal Neuropathy (GAN) causes a shortage of functional Gigaxonin. Nerves stop working normally in people with GAN. This causes problems with walking and sometimes with eating, breathing, and many other activities. GAN has no cure. Over time, GAN can shorten a person s life. Researchers want to see if a gene transfer treatment may help people with GAN.

Objectives:

- To see if a gene transfer is safe and shows potential to help people with GAN.

Eligibility:

- People age 3 and older with GAN.

Design:

* For 1 month following gene transfer participants must live full-time within 100 miles of the NIH.
* Participants will be screened by phone and in person. They will take many tests. Some are listed below. Their medical records will be reviewed. Their caregivers may be contacted.
* Participants will have a total of about 27 visits, weekly, monthly, and then yearly over 15 years. They will include many of the tests below.
* Physical and nervous system exams.
* Blood, urine, and stool samples.
* Nerve, lung, heart, and eye tests.
* Questionnaires.
* MRI scans, nerve biopsies, and spinal taps. Participants will be sedated for some tests.
* Speech, memory, muscle, and mobility tests.
* Skin biopsy (small sample removed).
* Participants will take many medicines. Some require intravenous lines.
* Participants will get the gene transfer through an injection by spinal tap into their cerebrospinal fluid, which flows around the brain and spinal cord. The genes are packed in a modified virus that carries the genes to cells in their body. Participants safety is not guaranteed.

DETAILED DESCRIPTION:
This is an open-label and non-randomized first-in-human (Phase 1) clinical trial which incorporates an escalating single dose paradigm to assess safety of the gene transfer vector scAAV9/JeT-GAN administered intrathecally to target the brain and spinal cord of individuals with genetically confirmed Giant Axonal Neuropathy (GAN, OMIM #256850).

GAN is a chronic neurodegenerative autosomal recessive disease pathologically characterized by enlarged axons with disordered intermediate filaments and microtubules. The disease pathology is due to loss-of-function variants in the GAN gene, which encodes the protein gigaxonin. Gigaxonin plays a major role in the maintenance of orderly and functional intermediate filament (IF) architecture, which is critical for axonal function. Onset of symptoms, usually at three to four years of age, generally manifests with a clumsy and unsteady gait (sensory ataxia). In the peripheral nervous system, the disease progressively affects predominantly sensory and motor nerves. By the end of the second decade of life, patients typically are wheelchair dependent with limited use of the arms and little to no use of their legs. During the second decade a tracheostomy or other means of ventilation, as well as a feeding tube, are often necessary. Death normally occurs in the second or third decade of life. We recently identified a sub-cohort of patients with a milder and later onset, yet progressive form of GAN characterized by a prolonged preservation of ambulation and less extensive white matter changes on brain MRI restricted to the infratentorial regions. These individuals are good trial candidates given the increased prospect of benefit at milder disease stages. There are no statistics on the incidence of GAN, but it is considered extremely rare and does not have an approved treatment aside from supportive care. Intrathecal delivery of a gene transfer vector carrying a normal copy of the GAN to the spinal cord and brain offers a potentially effective treatment for GAN.

Primary objective: To assess the safety of scAAV9/JeT-GAN following intrathecal administration.

Primary endpoint: Incidence of SAEs and treatment emergent adverse events at least possibly related to scAAV9/JeT-GAN treatment.

Secondary objectives:

1. to assess motor and sensory disease symptoms pre- and post-treatment,
2. to examine neuropathology in peripheral nerve biopsies in response to treatment,
3. to examine cerebrospinal fluid (CSF) and to conduct CSF studies to assess response to treatment, and
4. to assess vector shedding following vector administration.

Secondary endpoints: include clinical and physiological assessment of motor and sensory function, possible rescue of disease pathology in peripheral nerves, examination of CSF in response to treatment, and assessment of vector shedding following administration. The primary efficacy endpoint is the Motor Function Measure 32 (MFM-32).

Summary of progress through protocol version 23

A total of 14 trial participants (all >= five years of age) have received a single dose of scAAV9/JeTGAN ranging from 3.5 x 10^13 vg (1x dose) to 3.5 x10^14 vg (10x dose). Dosed individuals include those predicted to be cross-reactive immunological material (CRIM) positive (residual gigaxonin expression, n= 10) or CRIM-negative (absence of gigaxonin expression, n= 4), based on their respective GAN variant(s). In CRIM-positive individuals, residual protein expression may allow for transgene immune tolerance whereas in CRIM-negative individuals, immune modulation is required. Since GAN is a progressive neurodegenerative condition, younger and milder affected individuals have a higher prospect of benefitting from treatment with scAAV9/JeT-GAN. The study will explore the safety and efficacy in up to 21 patients with GAN ages 3 years and older, with an emphasis on enrollment of patients who are younger or with a

milder phenotype and are independently ambulant.

ELIGIBILITY:
* INCLUSION CRITERIA:

To participate in this study, subjects must meet the following criteria:

* Age 3 years or older.
* Genetic diagnosis of GAN: Identified pathogenic variant(s) on both copies of the GAN gene. If the variants found are not previously reported, then predictive software tools will be utilized to determine the degree of certainty that the variant is expected to be pathogenic (disease causing). This will also be evaluated in the context of the clinical and pathological phenotype.
* Men capable of fathering a child must agree to use barrier contraception (combination of a condom and spermicide) or limit activity to post-menopausal, surgically sterilized, or contraception-practicing partners, for 6 months after administration of investigational product. Women and girls of childbearing potential (and parents/ guardians for minors < 18) must agree to have urine human chorionic gonadotropin testing performed to rule out the possibility of pregnancy at each visit. Those women who are sexually active must also agree to use barrier contraception as well or limit activity to surgically sterilized or contraception-practicing partners for 3-6 months after the administration of the investigational product. This limitation is set because of the unknown risk associated with the administration of this vector genome to offspring. There is no known risk of sexual transmission of the vector.
* Willing and able to give informed consent if >17 years of age and assent if >7 years of age. For patients ages 7-17, parents or legal guardians must also consent to the child s participation in the study. Adults who lack capacity to consent but who have an appropriate surrogate may be included.
* Willingness to undergo a nerve biopsy at baseline and at 12 months after treatment.
* Agree to reside within 100 miles of the study site for at least 4 weeks following treatment (may include housing on NIH campus).

EXCLUSION/DEFERRAL CRITERIA:

To participate in this study, a patient MUST NOT have the following characteristics:

* Pregnant or lactating patients
* Forced vital capacity <= 50% of predicted value (if patient is >/= 5 years old; otherwise, baseline FVC is not required in those < 5 years old at time of enrollment)
* Ventilator dependence to include daytime use of assisted ventilation
* Current clinically significant infections including any requiring systemic treatment including but not limited to Human immunodeficiency virus, Hepatitis A, B, or C, Varicella zoster virus, or HTLV-1
* Prior history of bacterial meningitis
* Unwilling to undergo lumbar puncture at baseline and up to 2 to 3 times during follow up during the first year after treatment.
* Clinically significant echocardiogram abnormality per PI, anesthesiologist, and cardiologist
* Clinically significant electrocardiogram (ECG) abnormality per PI, anesthesiologist, and cardiologist
* History of brain or spinal cord disease that would interfere with the LP procedures, CSF circulation, or safety assessments
* Presence of an implanted shunt for the drainage of CSF or an implanted CNS catheter
* Any prior participation in a study in which a gene therapy vector or stem cell transplantation was administered to avoid any ambiguity in the safety assessment resulting from lingering effects from a previous treatment.
* Participation in an IND, IDE, or equivalent clinical study in the past six months.
* History of or current chemotherapy, radiotherapy or other immunosuppressive therapy within the past 30 days. Corticosteroid treatment may be permitted at the discretion of the PI.
* Immunizations of any kind in the month prior to the study to avoid lingering immune effects that could be confusing in the safety assessment of the trial.
* Current use of medication (e.g., levothyroxine, vitamin A supplementation, oral contraceptive use, tetracycline, Diamox etc) that could potentially lead to changes in intracranial pressure
* Known sensitivity or adverse reaction to anesthetic medications likely to be used in the peri-operative period per the anesthesiologist s evaluation
* GAN subjects without quantifiable weakness or functional loss
* Evidence of cardiomyopathy on history, exam, or additional testing (echocardiogram or electrocardiogram) or other cardiac disease that in the opinion of the investigator would deem the subject unsafe to participate in the trial
* History of diabetes or clinically significant abnormality of glucose tolerance test, fasting blood sugar
* Positive purified protein derivative testing for tuberculosis
* Abnormal laboratory values considered clinically significant per the investigator:

  * Platelet count < 100,000 / mm3
  * Persistent leukopenia or leukocytosis (Total white blood cell count < 3,000/mm and > 12,000/mm respectively)
  * Significant anemia [Hb <10 g/dL]
  * Abnormal prothrombin (PT) or partial thromboplastin time (PTT) [value]
  * Abnormal liver function tests (>1.5 X ULN or > 2 X the baseline value)
  * Abnormal pancreatic enzymes (>1.5 X ULN or > 2 X the baseline value)
  * Patients with renal impairment defined as urinary protein concentration >= 0.2 g/L on 2 consecutive tests
* Failure to thrive, defined as:
* Falling 20 percentiles (20/100) in body weight in the 3 months preceding Screening/Baseline
* In patients below the 3rd percentile, any further drop in body weight percentile in the 3 months preceding Screening/Baseline
* Weight less than < 3rd percentile predicted for age and gender based upon WHO criteria
* Any anticipated need for major surgery in the next 12 - 18 months (including scoliosis correction surgery)
* Ongoing medical condition that is deemed by the Principal Investigator to interfere with the conduct or assessments of the study

Ages: 3 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2015-04-24 (Actual); Primary Completion 2030-06-30 (Estimated); Study Completion 2035-04-01 (Estimated)

PRIMARY OUTCOMES:
To assess the safety of the vector | 12 months
  Adverse event reports will be used to assess safety

SECONDARY OUTCOMES:
Assessment of motor and sensory disease symptoms compare to baseline | 12 months
  Physical therapy assessments will be used for motor symptoms. Nerve conduction studies will be used to assess sensory symptoms.
Examination of neuropathology in peripheral nerve biopsies following treatment | 12 months
  Nerve biopsies will be collected and analyzed to examine neuropathology.
Examination of cerebrospinal fluid following treatment | 12 months
  CSF will be collected via lumbar puncture and analyzed to monitor for inflammatory markers.
Assessment of vector shedding following treatment | 12 months
  Biospecimens will be collected to analyze vector shedding.
Determine safety and tolerability of gene transfer in patients with null mutations receiving immunosuppression | 12 months
  Adverse event reporting will be used to assess the safety of gene transfer in CRIM-negative patients.

CONTACTS AND LOCATIONS:
Overall Officials: Carsten G Bonnemann, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All subject level data collected as part of the clinical trial will be shared. A CTA has been executed.
Supporting Information: Study Protocol
Time Frame: At a minimum, the study protocol will be shared with a commercial partner to assist with the BLA. The current CTA requires sharing of data by the end of July 2021; however, there are plans to extend the agreement until July 2023.
Access Criteria: A relationship has been established with a Taysha Gene Therapies. A data analysis plan has not yet been established by the company because NINDS is the current Sponsor.@@@@@@Safety is the primary outcome measure for this clinical trial.

REFERENCES:
- [Derived] Bharucha-Goebel DX, Todd JJ, Saade D, Norato G, Jain M, Lehky T, Bailey RM, Chichester JA, Calcedo R, Armao D, Foley AR, Mohassel P, Tesfaye E, Carlin BP, Seremula B, Waite M, Zein WM, Huryn LA, Crawford TO, Sumner CJ, Hoke A, Heiss JD, Charnas L, Hooper JE, Bouldin TW, Kang EM, Rybin D, Gray SJ, Bonnemann CG; GAN Trial Team. Intrathecal Gene Therapy for Giant Axonal Neuropathy. N Engl J Med. 2024 Mar 21;390(12):1092-1104. doi: 10.1056/NEJMoa2307952. PMID 38507752
- [Derived] Armao D, Bouldin TW, Bailey RM, Gray SJ. Extensive rod and cone photoreceptor-cell degeneration in rat models of giant axonal neuropathy: implications for gene therapy of human disease. Ophthalmic Genet. 2021 Oct;42(5):600-603. doi: 10.1080/13816810.2021.1923036. Epub 2021 May 6. PMID 33955818
- [Derived] Armao D, Bouldin TW, Bailey RM, Hooper JE, Bharucha DX, Gray SJ. Advancing the pathologic phenotype of giant axonal neuropathy: early involvement of the ocular lens. Orphanet J Rare Dis. 2019 Feb 1;14(1):27. doi: 10.1186/s13023-018-0957-5. PMID 30709364
- [Derived] Bailey RM, Armao D, Nagabhushan Kalburgi S, Gray SJ. Development of Intrathecal AAV9 Gene Therapy for Giant Axonal Neuropathy. Mol Ther Methods Clin Dev. 2018 Feb 15;9:160-171. doi: 10.1016/j.omtm.2018.02.005. eCollection 2018 Jun 15. PMID 29766026
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2015-N-0073.html